CLINICAL TRIAL: NCT05292742
Title: A Randomized, Open-label, Multicenter Study Comparing Continuation of Original Targeted Therapy With Trastuzumab Combined With Pyrotinib and Capecitabine as Postoperative Adjuvant Therapy in Non-pCR Patients With HER2 Positive Early Breast Cancer
Brief Title: Compare Continuation of Original Targeted Therapy With Trastuzumab Combined With Pyrotinib and Capecitabine as Postoperative Adjuvant Therapy in Non-pCR Patients With HER2 Positive Early Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-025
Record Dates: First submitted 2022-02-23; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer; Adjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Pyrotinib: 400 mg/day (once daily, orally at the same time every day), every 3 weeks for one year Capecitabine: 1000 mg/m2 orally twice daily every 3 weeks for 6 cycles Trastuzumab: Initial loading dose of 8 mg/kg followed by 6 mg/kg every 3 weeks. One year of trastuzumab treatment (including: neoadjuvant phase and adjuvant phase)
  Interventions: Drug: Pyrotinib+Trastuzumab+Capecitabine
- B (Active Comparator): Patients in the control group will continue neoadjuvant targeted therapy, trastuzumab or trastuzumab in combination with pertuzumab. In case of neoadjuvant trastuzumab monotherapy, trastuzumab combined with pertuzumab targeted therapy is allowed in the adjuvant phase.
  Interventions: Drug: Trastuzumab+Pertuzumab/Trastuzumab

INTERVENTIONS:
Drug: Pyrotinib+Trastuzumab+Capecitabine — Patients in the experimental arm will receive trastuzumab + pyrotinib + capecitabine
  Arms: A
Drug: Trastuzumab+Pertuzumab/Trastuzumab — Trastuzumab: Initial loading dose of 8 mg/kg followed by 6 mg/kg every 3 weeks. One year of trastuzumab treatment (including: neoadjuvant phase and adjuvant phase) Pertuzumab: 840 mg loading dose followed by 420 mg fixed dose
  Arms: B

SUMMARY:
To evaluate the efficacy of continuation targeted therapy compared with trastuzumab combined with Pyrotinib and capecitabine in postoperative adjuvant therapy of HER-2 positive early breast cancer patients with residual tumor (primary breast tumor/axillary lymph nodes) who did not achieve pCR after neoadjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 years and ≤ 75 years old with primary breast cancer
* ECOG score 0 ~ 1
* Breast cancer meets the following criteria: 1）Histologically or pathologically confirmed invasive breast cancer, primary tumor stage determined by standard evaluation methods：cT1-4/N0-3/M0. 2）Pathologically confirmed HER2-expressing positive breast cancer, defined as > 10% immunoreactive cells with immunohistochemical (IHC) score of 3 + or in situ hybridization (ISH) results of HER2 gene amplification. 3)Known hormone receptor status (ER and PgR). 4)Neoadjuvant therapy (including: at least 9 weeks of trastuzumab treatment and at least 9 weeks of taxane chemotherapy)
* Primary breast cancer lesion or lymph node invasive cancer confirmed by pathology after neoadjuvant therapy (residual invasive breast cancer lesion > 2 cm or axillary lymph node positive with macrometastasis assessed by central laboratory)
* No more than 12 weeks between end of surgery (without post-operative radiotherapy) and randomisation or 6 weeks between end of post-operative radiotherapy and randomisation
* Required laboratory values including following parameters:

ANC: ≥ 1.5 x 109/L Platelet count: ≥ 90 x 109/L Hemoglobin: ≥ 9.0 g/dL Total bilirubin: ≤ 1.5 x upper limit of normal, ULN ALT and AST: ≤ 1.5 x ULN BUN and creatine clearance rate: ≥ 50 mL/min LVEF: ≥ 55% QTcF: < 470 ms

Exclusion Criteria:

* 1) Stage IV (metastatic) breast cancer;
* 2) inflammatory breast cancer;
* 3) Previous anti-tumor therapy or radiotherapy for any malignancy, excluding cured cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma;
* 4) Receiving anti-tumor therapy in other clinical trials, including bisphosphonate therapy or immunotherapy (except radiotherapy and endocrine therapy during treatment);
* 5) Receiving any anti-tumor therapy within 28 days before enrollment;
* 6) Peripheral neuropathy ≥ Grade 2 as specified by NCI CTCAE;
* 7) Receiving pyrrolidone or other anti-HER2 tyrosine kinase inhibitors;
* 8) Receiving anthracycline therapy with cumulative doses as follows: adriamycin > 240 mg/m2, epirubicin > 480 mg/m2;
* 9) Receiving major surgery unrelated to breast cancer before randomization, or the patient has not fully recovered from surgery

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
iDFS | 3 years
  3-year invasive disease-free survival (iDFS) rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China